CLINICAL TRIAL: NCT05274867
Title: Development of a Patient Reported Outcome Measure for Advanced Ovarian Cancer Patients Receiving Surgical and Chemotherapy Treatment
Acronym: PROM-OSP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp208
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer; Surgery; Chemotherapy; Patient Reported Outcome Measure
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development of a patient reported outcome measure (PROM) for ovarian cancer patients receiving combined surgery and radiotherapy

DETAILED DESCRIPTION:
The study will be conducted in four stages:

Stage I - Item generation Approximately 20 interviews will be conducted with ovarian patients receiving combined surgery and chemotherapy to capture their experiences including quality of life, symptom experience, and other relevant themes that may emerge. The interviews will be audio recorded and transcribed verbatim. The qualitative data will be analysed thematically and key quotes extracted which will be used to create a draft item list. Interviews will be conducted either in person or virtually depending on national social distancing guidance at the time. Interviews will be audio recorded using a Dictaphone which encrypts files in real time.

Stage II - Cognitive interviewing Following the initial interviews, approximately 7 participants will undergo cognitive interviews to ensure that all items are clear and easily understood. Interviews will be audio recorded using a Dictaphone which encrypts files in real time.

Stage III - Item reduction and refinement of the draft PROM A draft PROM and the EORTC QLQ-C30 (a validated measure of health related quality of life for cancer patients in clinical trials) will be administered to approximately 100 ovarian cancer participants receiving combined surgery and chemotherapy. Approximately 50 patients will be asked to repeat the draft PROM approximately one week later to assess test-retest reliability. Hierarchical item reduction and Rasch analysis will be used to determine which items should be included in the final PROM.

Stage IV- Pilot testing The final PROM will be pilot tested with approximately 10 patients at The Christie site to assess its acceptability

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving combined surgery and chemotherapy for advanced ovarian cancer
* Aged over 18 (no upper age limit)
* Ability to understand and communicate in the English language
* Able to provide written informed consent

Exclusion Criteria:

* Patients who are not receiving combined surgery and chemotherapy for advanced ovarian cancer
* Unable to understand and communicate in the English language
* Aged under 18
* Unable to provide written informed consent
* Patients who are not able to complete informed consent or the study questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women receiving combined surgery and chemotherapy treatment for advanced ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-06-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
European Organisation Research and Treatment of Cancer Quality of Life- Core 30 (EORTC | 4 weeks
  Generic cancer quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sally Taylor, PhD, Principal Investigator — The Christie NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No